CLINICAL TRIAL: NCT06219863
Title: Feasibility and Outcome Measures for Infants With Down Syndrome: Advancing Clinical Trial Readiness for a Harness-based Mobility Intervention
Brief Title: Harness-based Mobility Intervention for Infants With Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Jana M. Iverson, Christopher A. Moore Professor of Pediatric Rehabilitation, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6930E
Record Dates: First submitted 2023-12-30; First posted 2024-01-23 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Down Syndrome
Keywords: infant
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Body weight supported harness (Experimental): Harness is set up in families' homes for one month. Caregivers re asked to use the harness with their infant for 30 min/day, 5 times a week.
  Interventions: Behavioral: Body weight supported harness

INTERVENTIONS:
Behavioral: Body weight supported harness — A body weight supported harness will be provided to families for one month to set up in their home. Caregivers will be asked to use the harness for their infants for 30 min per day, 5 days a week. Caregivers will complete a daily log describing harness use. At the end of the month, they will complete feasibility and acceptability questionnaires.

SUMMARY:
The emergence of crawling and walking is significantly delayed in infants with Down syndrome (DS), but the development of independent mobility provides infants with new opportunities for exploring the environment and interacting with objects and people that are important foundations for early learning. Increasing infant mobility early in development with body weight supported harness systems may support infant exploration, communication, and social interaction. This project will set the stage for the first clinical trial of a mobility-related intervention specifically tailored for infants with DS by testing the feasibility of harness systems with infants and families and identifying measures that will serve as primary outcome variables. Upon completion of this pilot project, necessary preliminary data and experience required for an in-home, high-impact clinical trial for infants with DS will have been obtained.

DETAILED DESCRIPTION:
Investigators will visit families at home both in-person and virtually via Zoom. At all sessions, infants and caregivers will be videorecorded at home while playing together with the infant's own toys (15 min) and with a standard set of age-appropriate commercially available toys provided by the research team (15 min). During the harness trial period, sessions will be divided so that the infant is observed both in and out of the harness. Parent reports of language development (MacArthur-Bates Communicative Development Inventory; 10 min) and locomotor development (Locomotor Experience Interview; 10 min) will be collected at the initial visit, study midpoint (3 months), and study exit (6 months). Parents will be surveyed once about the feasibility and acceptability of the body weight supported harness system at the end of the harness trial period (10 min), and they will complete a study participation satisfaction survey at study exit (10 min). In addition, infants will be administered the Bayley Scales of Infant and Toddler Development-4 (30 min) and the Early Social Communication Scales (10 min) at the beginning, middle, and end of study participation.

Participants will be observed twice a month for 6 months (one visit per month on Zoom and the other in person), for a total of 12 observations per child.

Part 2 study participation will involve a total of 12 sessions per parent/infant dyad, lasting between 30 and 70 min, depending on the visit protocol (see above).

Each family will also have a 1-month Harness Trial Period with the PUMA system in their home. These will be staggered over the course of the study period. At the beginning of the trial period, investigators will deliver the harness system to the home and assist with setup and troubleshooting. Families will be given a brief training in harness setup and use and a safety checklist to review daily before using the system with their infant. Families will be asked to use the harness with their infant for at least 30 minutes daily. The harness will be collected by the research team at the end of the trial period. Each day during the Harness Trial Period, parents will track how long they use the harness system with their infant (in minutes), what activities they engaged in (e.g., toy play, book sharing), and any challenges they encountered (e.g., infant fussiness) in a log (5 min).

The PUMA system is an FDA registered device manufactured by Enliten LLC that provides body weight support while moving around. It consists of a 9' x 9' metal canopy frame with no cover that is adjustable in height. Infants will wear custom lightweight cloth vests designed specifically for the PUMA. The vest will be connected to a beam at the top of the structure. The PUMA supports up to 60 pounds and permits movement anywhere beneath the structure. In case of an emergency, a quick release unit can be pulled to rapidly separate the harness from the support unit. For the PUMA, this device is attached to the spreader bar, out of reach of the child user.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Trisomy 21
* younger than 24 months
* English is the primary language of the home (due to use of standardized language assessments normed on English-speaking children)
* able to sit without support
* not yet taking any independent steps.

Exclusion Criteria:

* Mosaic or Translocation Down syndrome
* severe, uncontrolled medical problems (including heart disease with cardiovascular instability, uncontrolled epilepsy)
* severe uncorrected hearing or vision impairments

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean posture duration in seconds | 6 months
  Average time spent in supine, prone, sitting, standing
Mean number of locomotion bouts | 6 months
  Mean instances of crawling, cruising, walking, or other forms of locomotion
Mean time spent in contact with objects | 6 months
  Average time infants spend touching objects
Mean number of different objects contacted | 6 months
  Average number of unique objects touched
Mean number of vocalizations | 6 months
  Average number of speech-like sound productions
Mean number of gestures | 6 months
  Average number of gestures
Proportion of directed vocalizations | 6 months
  Proportion of total vocalizations accompanied by looking to the caregiver
Proportion of directed gestures | 6 months
  Proportion of total gestures accompanied by looking to the caregiver
Bayley Scales of Infant Development-4 | Study entry, 3 months, 6 months
  Comprehensive, standardized measure of general development for children from 1-42 months, with five subscales: Cognitive, Language, Motor, Social-Emotional, and Adaptive Behavior. Raw scores will be used. Minimum score is 0; there is no maximum score. Higher scores indicate a better outcome.
Early Social Communication Scales | Study entry, 3 months, 6 months
  Structured experimenter-administered observation of nonverbal communication skills: assesses joint attention, requesting, and social interaction skills. Minimum score is 0. There is no maximum score. Higher scores mean a better outcome.
MacArthur-Bates Communication Development Inventory: Words & Gestures | Study entry, 3 months, 6 months
  Parent questionnaire identifying words that the child only understands and those that s/he both says and understands as well as production of early gestures (e.g., showing, pointing) and actions (e.g., games, routines). There are seven subscales. Raw scores will be reported for each one, and all have a minimum score of 0. Higher scores mean better outcomes.
  Words Understood (maximum score = 396) Words Produced (maximum score = 396) First Communicative Gestures (maximum score = 12) Games and Routines (maximum score = 6) Actions with Objects (maximum score = 17) Pretending to be a Parent (maximum score = 13) Imitating Other Adult Actions (maximum score = 15)

CONTACTS AND LOCATIONS:
Overall Officials: Jana Iverson, PhD, Principal Investigator — Boston University; Nicole Baumer, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from standardized assessments will be shared with the NIH INCLUDE database.
Time Frame: One year after study completion
Access Criteria: Access granted to approved users of the INCLUDE database